CLINICAL TRIAL: NCT04270630
Title: A Pilot Proof of Concept, Randomized Controlled, Single-Center Study of a Decision Aid Tool for Older Patients (Age ≥75) Considering Left Heart Catheterization as Treatment for Non-St Elevation Myocardial Infarction
Brief Title: A Pilot Proof of Concept, Randomized Controlled, Single-Center Study of a Decision Aid Tool for Older Patients Considering LHC as Treatment for NSTEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-01687
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: NSTEMI
Keywords: Shared decision making; Left heart catheterization; Non-ST elevation myocardial infarction; Decisional conflict; Decision aid
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Patients in the control arm of the study will undergo standard of care treatment, discussing catheterization with their treating physicians.
- Shared decision aid (Experimental): Patients in the interventional arm of the study will discuss catheterization with their treating physicians, in addition to having access to the shared decision aid tool and a shared decision conversation with a co-investigator clinician.
  Interventions: Behavioral: Shared Decision Aid

INTERVENTIONS:
Behavioral: Shared Decision Aid — The decision aid was developed by this study group based on the International Patient Decision Aid Standards Collaboration's minimum standards for quality, and the Ottawa Framework (a process by which patients' and clinicians' decision determinants are assessed, a decision aid is developed that is tailored to these needs, and the quality of the decision-making process with the aid is evaluated). The aid then underwent an iterative feedback process with a patient advisory panel. Adjustments to format, length, and readability were made. A final feedback session occurred with three patients over the age of 70, after which point the paper decision aid was digitalized. The intervention will be delivered in-person by one of the co-investigators of the study. The intervention will occur once, prior to the patient making a final decision regarding undergoing left heart catheterization as treatment for NSTEMI. The approximate duration of the intervention is 30 minutes.
  Arms: Shared decision aid

SUMMARY:
This study will be a single-center, prospective, un-blinded, randomized controlled trial evaluating a decision aid tool for older patients considering left heart catheterization (LHC) as treatment for non-ST elevation myocardial infarction (NSTEMI). The study population is 50 total inpatients (25 per study arm) with NSTEMI eligible for elective LHC. The first arm is the control group that will receive standard of care, while the second arm will have access to the decision aid and shared-decision making conversation with one of the co-investigators. Baseline characteristics and surveys/questionnaire data will be collected after study intervention (as applicable), and prior to final decision regarding LHC. Statistical analyses will be conducted on the primary endpoint, decisional conflict score, as well as on various secondary endpoints.

DETAILED DESCRIPTION:
A single-center, prospective, un-blinded, randomized controlled trial. Primary objective: To pilot a coronary revascularization decision aid in older adults with NSTEMI who are candidates for elective LHC in order to determine its effectiveness in lowering decisional conflict by the decisional conflict scale (DCS).

Secondary objectives: To determine decision aid feasibility by measuring time of administration and percentage of patients agreeing to use. Also, to assess efficacy of the decision aid in decreasing patient feelings of anxiety and depression (by the Hospital Anxiety and Depression Scale), increasing decision self-efficacy (by the Ottawa Decision Self-Efficacy Scale), and increasing medical knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Must be admitted to the hospital, and there must be clinical suspicion for type I NSTEMI
* Must be eligible for non-urgent revascularization
* Must have capacity to consent for the study based on the judgment of the study investigators
* Must speak English

Exclusion Criteria:

* Does not meet all of the inclusion criteria listed above
* Has significant vision or hearing impairment that prohibits use of the decision aid
* Unable to read
* Has a clinical diagnosis of dementia and/or severe cognitive impairment documented in the electronic medical record

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Percent change in mean decisional conflict score between the control and interventional group | Visit 1 (Day 0)
  A reduction in decisional conflict score will be measured with the DCS tool to reflect an increase in the quality of the decision.

SECONDARY OUTCOMES:
Descriptive Statistics in the use of the Patient Decision Aid | Visit 1 (Day 0)
  Descriptive differences in the participants who use the patient decision aid and those who are in the control group will be measured with study surveys

CONTACTS AND LOCATIONS:
Overall Officials: John Dodson, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to rachel.sibley@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.